CLINICAL TRIAL: NCT01343966
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel-Group, Multicenter, Phase II Study to Evaluate the Efficacy and Safety of MABT5102A in Patients With Mild to Moderate Alzheimer's Disease (ABBY)
Brief Title: A Study to Evaluate the Efficacy and Safety of MABT5102A in Patients With Mild to Moderate Alzheimer's Disease (ABBY)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABE4869g; ABBY (Other: Genentech); GN00761 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2011-04-27; First posted 2011-04-28 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-07

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — crenezumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Part 1: Subcutaneous cohort exp (Experimental)
  Interventions: Drug: MABT5102A
- Part 2: Intravenous cohort exp (Experimental)
  Interventions: Drug: MABT5102A
- Part 1: Subcutaneous cohort (Placebo Comparator): Repeating subcutaneous injection
  Interventions: Drug: placebo
- Part 2: Intravenous cohort (Placebo Comparator): Repeating intravenous infusion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: MABT5102A — Repeating subcutaneous injection
  Arms: Part 1: Subcutaneous cohort exp
Drug: MABT5102A — Repeating intravenous infusion
  Arms: Part 2: Intravenous cohort exp
Drug: placebo — Repeating subcutaneous injection
  Arms: Part 1: Subcutaneous cohort
Drug: placebo — Repeating intravenous infusion
  Arms: Part 2: Intravenous cohort

SUMMARY:
This is a Phase II, randomized, double-blind, parallel-group, placebo-controlled study to evaluate the safety and efficacy of MABT5102A in patients with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable AD according to the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorder Association (NINCDS-ADRDA) criteria
* Mini-Mental State Examination (MMSE) score of 18-26 points at screening
* Geriatric Depression Scale (GDS-15) score of < 6
* Completion of 6 years of education (or good work history consistent with exclusion of mental retardation or other pervasive developmental disorders)
* If receiving concurrent AD treatment, patient must be on the medication for at least 3 months at a stable dose for at least 2 months prior to randomization.

Exclusion Criteria:

* Severe or unstable medical condition that, in the opinion of the investigator or Sponsor, would interfere with the patient's ability to complete the study assessments or would require the equivalent of institutional or hospital care
* History or presence of clinically evident vascular disease potentially affecting the brain
* History of severe, clinically significant (persistent neurologic deficit or structural brain damage) central nervous system trauma
* Hospitalization within 4 weeks prior to screening
* Previous treatment with MABT5102A or any other therapeutic that targets Abeta
* Treatment with any biologic therapy within 5 half-lives or 3 months prior to screening, whichever is longer, with the exception of routinely recommended vaccinations, which are allowed

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2011-04-30 (Actual); Primary Completion 2014-02-28 (Actual); Study Completion 2014-02-28 (Actual)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale Cognitive Subscale (ADAS-Cog) score | From baseline to Week 73
Change in Clinical Dementia Rating, Sum of Boxes (CDR-SOB) score | From baseline to Week 73

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) score | From baseline to Week 73

CONTACTS AND LOCATIONS:
Overall Officials: Robert Paul, M.D., Ph.D., Study Director — Genentech, Inc.
Locations (92):
- United States (40):
  - Hope Research Institute, Phoenix, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Pharmacology Research Inst, Encino, California
  - Margolin Brain Institute, Fresno, California
  - Univ of CA San Diego; Neurosciences Comp.Alzheimer's, La Jolla, California
  - USC School of Medicine, Los Angeles, California
  - Pharmacology Research Inst, Newport Beach, California
  - University of California Davis Medical System, Sacramento, California
  - Pacific Research Network - PRN, San Diego, California
  - Uni of California San Francisco, San Francisco, California
  - Neurological Research Inst, Santa Monica, California
  - Yale University, New Haven, Connecticut
  - Florida Atlantic University; College of Medicine, Boca Raton, Florida
  - Meridien Research, Brooksville, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Miami Jewish Health Systems; Clinical Research, Miami, Florida
  - Collier Neurologic Specialists, Naples, Florida
  - Compass Research, Orlando, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Rush Alzheimer's Disease Cntr., Chicago, Illinois
  - Alexian Brothers Neurosci Inst, Elk Grove Village, Illinois
  - IU Healthy Partners Adult Neurology Clinic, Indianapolis, Indiana
  - Louisiana Research Associates, New Orleans, Louisiana
  - Millennium Psychiatric Associates, LLC, Creve Coeur, Missouri
  - NeuroCognitive Institute, Mount Arlington, New Jersey
  - Memory Enhancement Center of NJ, Inc., Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - Empire Neurology, PC, Latham, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical Center; Monroe Community Hospital, Rochester, New York
  - Investigational Drug Service; Univ of Rochester Medical Ctr, Rochester, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Neurology & Neuroscience Ctr of Ohio, Toledo, Ohio
  - Clinical Trials of America, Inc., Eugene, Oregon
  - Summit Research Network Inc., Portland, Oregon
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Medical Uni of South Carolina, North Charleston, South Carolina
  - Alzheimers Disease & Memory Disorders Center; Department of Neurology Baylor College of Medicine, Houston, Texas
  - Clinical Neuroscience Research Associates, Inc., Bennington, Vermont
- Canada (16):
  - Saibal Nandy Professional Corporation, Medicine Hat, Alberta
  - The Med Arts Health Rsrch Grp, Kelowna, British Columbia
  - The Med Arts Health Rsrch Grp, Penticton, British Columbia
  - University of British Columbia Hospital; Division of Neurology, Vancouver, British Columbia
  - Capitol District Health Authority, Halilfax, Nova Scotia
  - Jbn Medical Diagnostic Services Inc., Burlington, Ontario
  - Hotel Dieu Hospital, Kingston, Ontario
  - Providence Care Centre; Mental Health Site, Kingston, Ontario
  - St. Joseph's HC-Parkwood Hosp, London, Ontario
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Regional Memory Clinic, Peterborough, Ontario
  - Toronto Memory Program (Neurology Research Inc.), Toronto, Ontario
  - Clinique Neuro Rive-Sud, Greenfield Park, Quebec
  - Hôpital Maisonneuve-Rosemont/Polyclinique;Recherche Clinique, Montreal, Quebec
  - CHAUQ Hopital Enfant-Jesus, Québec, Quebec
  - McGill Univeristy; Douglas Mental Health University Institute; Neurological and Psychiatric, Verdun, Quebec
- France (9):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital neurologique Pierre Wertheimer - CHU Lyon; Neurologie, Bron
  - Chu Limoges, Limoges
  - Hopital Nord Laennec, Nantes
  - Hopital de Cimiez, Nice
  - Hopital Broca, Paris
  - CHU de Rouen Hopital; Service de Neurologie, Rouen
  - Hopital Hautepierre; Centre dInvestigation Clinique, Strasbourg
  - Hôpital Casselardit; Cons memoire, Toulouse
- Germany (11):
  - Studienambulanz emovis GmbH; St. Joseph Krankenhaus, Berlin
  - Univ Berlin; Klin fur Psychi & Psycho Charite, Berlin
  - Universitätsklinikum Erlangen; Augenklinik, Erlangen
  - Bezirkskrankenhaus Günzburg, Günzburg
  - Zentralinstitut fuer Seelische Gesundheit, Mannheim
  - Inst fur Stedien zur Psych Ges, Mannheim
  - Psych Klin der LMU Muenchen, München
  - Ludwig-Maximilians-Univ., München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Villa Sauer, Praxis für; Neurologie und Psychiatrie, Siegen
  - Universitätsklinik Tübingen; Psychiatrie und Psychotherapie, Tübingen
- Spain (7):
  - Hospital General de Catalunya, San Cugat Del Valles, Barcelona
  - Policlinica Guipuzcoa, Donostia / San Sebastian, Guipuzcoa
  - Hospital de Cruces; Servicio de Neurologia, Barakaldo, Vizcaya
  - Hospital Perpetuo Socorro, Albacete
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Clinica Ruber, 4 planta; Servicio de Neurologia, Madrid
  - Hospital Universitario Virgen de la Macarena;, Seville
- United Kingdom (9):
  - The Rice Centre; Royal United Hospital, Bath
  - West London Research Unit; Brentford Lodge, Brentford
  - Royal Sussex County Hospital, CIRU Level 5, Brighton
  - Glasgow Memory Clinic, Glasgow
  - Camden Mews Day Hospital; Camden and Islington, London
  - The National Hospital for Neurology & Neurosurgery; Dementia Research Center, London, GT LON
  - Southampton General Hospital; Pharmacy, Southampton
  - Moorgreen Hospital; Memory Assessment & Rsch Ctr, Southampton
  - Great Western Hosp.; Kingshill Research Ctr, Swindon

REFERENCES:
- [Derived] Polhamus DG, Dolton MJ, Rogers JA, Honigberg L, Jin JY, Quartino A. Longitudinal Exposure-Response Modeling of Multiple Indicators of Alzheimer's Disease Progression. J Prev Alzheimers Dis. 2023;10(2):212-222. doi: 10.14283/jpad.2023.13. PMID 36946448
- [Derived] Yoshida K, Moein A, Bittner T, Ostrowitzki S, Lin H, Honigberg L, Jin JY, Quartino A. Pharmacokinetics and pharmacodynamic effect of crenezumab on plasma and cerebrospinal fluid beta-amyloid in patients with mild-to-moderate Alzheimer's disease. Alzheimers Res Ther. 2020 Jan 22;12(1):16. doi: 10.1186/s13195-020-0580-2. PMID 31969177